CLINICAL TRIAL: NCT04502420
Title: Hypoxia, Lung Function and Diffusion Capacity After Abdominal Surgery
Brief Title: Lung Function After Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Professor, Umeå University
Other Study IDs: 2018-223-31M
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Lung Function; Postoperative Complications; Abdominal Surgery
Keywords: Lung function; Diffusion capacity; Postoperative complications; Abdominal surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abdominal surgery: People who to be operated in the abdomen are investigated before and after surgery.
  Interventions: Diagnostic Test: Lung function before and after surgery

INTERVENTIONS:
Diagnostic Test: Lung function before and after surgery — A diagnostic test
  Other Names: Diffusion capacity and arterial blood gas before and after surgery.

SUMMARY:
The study aims to investigate changes in lung function and diffusion capacity for carbon monoxide after open and minimally invasive abdominal surgery and whether such changes can explain hypoxia after surgery.

Inclusion: Patients undergoing surgery for abdominal surgery

Exclusion: Dementia or cognitive impairment that makes it impossible to participate in studies.

Investigation: The day before surgery and the day after surgery

Primary outcome measures:

* Pulmonary function test with dynamic spirometry (Vital capacity, FEV1) and diffusion capacity for carbon monoxide.
* PaO2, PaCO2 and oxygen saturation (blood gas)

DETAILED DESCRIPTION:
Postoperative hypoxia complicates 30% - 50% of abdominal surgeries. People at particular risk for postoperative pulmonary complications including severe hypoxia are those who undergo abdominal surgery, emergency surgery or have a respiratory failure due to chronic lung disease including obstructive sleep apnea. The cause of postoperative restrictive lung function and hypoxia is unknown. Previous studies report that PaO2 decreases by an average of 2 kPa after abdominal surgery, while PaCO2 is unchanged and vital capacity decreases by 35%.

The study aims to investigate changes in lung function and diffusion capacity for carbon monoxide after open and minimally invasive abdominal surgery and whether such changes can explain hypoxia after surgery.

Design: Prospective cohort study

Inclusion: Patients undergoing surgery for abdominal surgery

Exclusion: Dementia or cognitive impairment that makes it impossible to participate in studies.

Method: The day before surgery and the day after surgery: Lung function (Vital capacity and FEV1) using box and diffusion capacity measurements and blood gas measurement

Primary outcome measures:

* Pulmonary function test with dynamic spirometry (Vital capacity, FEV1) and diffusion capacity for carbon monoxide.
* PaO2, PaCO2 and oxygen saturation (blood gas) Other variables examined: age, sex, height, weight, type of surgery, type of anesthesia, smoking status, length of surgery, previously known lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old and older) scheduled for surgery in the abdomen at department of Surgery, Urology and Gynecologi, Umeå University hospital.
* Must be able to perform a lung function test

Exclusion Criteria:

• Dementia or severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of 18 years old or olderundergoing abdominal surgery at department of Surgery, Urology and Gynecologi Umeå University hospital
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Diffusion capacity for carbon monoxide (DLCO) | Change from baseline (the day before surgery) to postoperative day 1 or 2
  Change in DLCO

SECONDARY OUTCOMES:
Vital capacity (VC) | Change from baseline (the day before surgery) to postoperative day 1 or 2
  Change in VC
Forced expiratory volume (FEV1) | Change from baseline (the day before surgery) to postoperative day 1 or 2
  Change in FEV1
Arterial PO2 | Change from baseline (the day before surgery) to postoperative day 1 or 2
  Change in arterial PO2
Arterial PCO2 | Change from baseline (the day before surgery) to postoperative day 1 or 2
  Change in arterial PCO2

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, Prof, Principal Investigator — Inst Surgical and periopertive sciences, Umeå university, Sweden
Locations (1):
- Dept surgery,, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
We plan to share IPD if possible according to Swedish legislation